CLINICAL TRIAL: NCT03878628
Title: Treatment With Allogeneic Adipose-derived Mesenchymal Stem Cells in Patients With Aqueous Deficient Dry Eye Disease
Acronym: MESADDE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Møller-Hansen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001-2018
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye; Kerato Conjunctivitis Sicca; Aqueous Tear Deficiency
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adipose tissue-derived mesenchymal stem cells (Experimental): Approximately 11 million ASCs in a 0.5 ml suspension
  Interventions: Drug: Adipose tissue-derived mesenchymal stem cells

INTERVENTIONS:
Drug: Adipose tissue-derived mesenchymal stem cells — CSCC_ASC(22), a ready-to-use suspension containing 22 million adipose tissue-derived mesenchymal stem cells per millilitre

SUMMARY:
The objective of this study is to assess the safety and feasibility of allogeneic adipose tissue-derived mesenchymal stem cells (ASCs) injected into the lacrimal gland in a smaller groups of 7 patients with Aqueous Deficient Dry Eye Disease (ADDE)

DETAILED DESCRIPTION:
Dry eye disease (DED) is a very common problem seen in patients all over the world. According to an older study the prevalence of DED in a Danish population 30-60 years of age was 11%. Aqueous tear deficient dry eye (ADDE) is a subtype of DED in which the tear production in the lacrimal gland (LG) is impaired. Current treatment of ADDE is only to relieve symptoms as a curative treatment of ADDE does not exist.

Mesenchymal stem cells (MSCs) reside in almost all connective tissues and are multipotent stem cells with the capacity to differentiate into several kinds of tissue. Several studies have shown that MSCs reduces inflammation in various diseases. Adipose tissue-derived MSCs (ASCs) have gained considerable attention, since they are readily available from the abdominal fat where it is most easily collected and expanded. In resting MSCs, MHC class II is not expressed on the surface, which reduces the inherent immunogenicity of the cells. This supreme attribute allows allogeneic MSC transplantation. Treatment with allogeneic MSCs have been investigated in an extensive number of human subjects for various conditions in clinical trials and no documented adverse events related to an anti-donor immune response exist. One potential advantage of treatment with allogeneic cells is the possibility of their use as an "off-the-shelf" therapeutic agent, avoiding the need for tissue collection and culture to delay and increase the cost of treatment. It has also been suggested that the function of autologous MSCs could be impaired in patients with comorbidities or advanced age.

In canines as in humans the most common cause of ADDE is an immune-mediated inflammatory response targeting the LG. Two studies with injection of allogeneic ASCs from healthy donors in a total of 48 eyes in 27 canines with ADDE have been performed with a significant increase in tear production and no observed adverse events to the treatment.

Studies with injection of ASCs into the human LG has never been conducted. This present study will test the hypothesis that injection of allogeneic ASCs into the LG in patients suffering from ADDE is safe and increases tear production and reduces inflammation resulting in increased ocular comfort.

7 patients with severe ADDE from Dept. of Ophthalmology, Rigshospitalet-Glostrup, will be recruited if they are 1: eligible for the study and 2: sign the informed consent form.

At inclusion the participants will fill out the Ocular Surface Disease Index (OSDI) questionnaire and undergo an eye examination in the following order:

measurement of tear osmolarity (TearLab™), tear break-up time (TBUT), ocular surface staining according to the Ocular SICCA Grading Score, and Schirmer's I test.

After a maximum of 14 days from screening all participants will receive an injection with ASCs into the lacrimal gland on one eye. If both eyes fulfill the eligibility criteria the most affected eye with the lowest tear production assessed with the Schirmer's I test will be the study eye; the contralateral eye will not be treated but examined according to the same protocol as the study eye at each follow-up.

The product used is CSCC_ASC(22) and the dose injected contains approximately 11 million ASCs per LG in a suspension with a total volume of 0.5 ml.

1 week (±2 days), 4 weeks (±4 days), and 4 months (±7 days) after intervention the participants are followed up with eye examination as described above, OSDI questionnaire, and blood test. At 4 months the primary outcomes of safety will be evaluated.

End of trial is defined as last participant's last visit (LPLV) at 3 years late follow-up.

ELIGIBILITY:
Inclusion Criteria:

* OSDI-score > 30
* Schirmer's test 2-5 mm in 5 minutes
* TBUT < 10 sec.

Exclusion Criteria:

* Previously established allergies to Oxybuprocaine or DMSO (rare)
* Reduced immune response (e.g. HIV positive)
* Pregnancy or planned pregnancy within the next 2 years
* Breastfeeding
* Treatment with an anticoagulant that cannot be stopped during the intervention period
* Treatment with systemic medication known to reduce tear production (with an odds ratio >2,0 (3)): anxiolytics, antipsychotics, and inhaled steroids.
* Topical treatment with eye drops other than lubricants
* Any other disease/condition judged by the investigator to be grounds for exclusion, such as infection in or around the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Pain at injection site: grade | 4 months after treatment
  grade 1: mild pain, grade 2: moderate pain, grade 3: severe pain
Infection at injection site | 4 months after treatment
  grade 1: localized; local intervention indicated, grade 2: oral intervention indicated (antibiotic, antifungal, antiviral), grade 3: intravenously administered (IV) antibiotic, antifungal, or antiviral agent indicated; or operative intervention indicated, grade 4: life-threatening consequences; urgent intervention needed.
Bleeding at injection site | 4 months after treatment
  Grade 1: Mild bleeding; intervention not indicated; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization indicated.
Eyelid function disorder | 4 months after treatment
  Grade 1: Asymptomatic; clinical or diagnostic observations only; intervention not indicated;
  Grade 2: Symptomatic; nonoperative intervention indicated; limiting instrumental ADL;
  Grade 3: Limiting self care ADL; operative intervention indicated.
Periorbital edema | 4 months after treatment
  Grade 1: Soft or non-pitting;
  Grade 2: Indurated or pitting edema; topical intervention indicated;
  Grade 3: Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated.
Ocular discomfort | 4 months after treatment
  grade 1: mild discomfort,
  grade 2: moderate pain,
  grade 3: disabling pain.
Flu-like symptoms | 4 months after treatment
  grade 1: Mild flu-like symptoms present;
  grade 2: Moderate flu-like symptoms, limiting self care ADL;
  grade 3: Severe flu-like symptoms, limiting self care ADL)
Fever | 4 months after treatment
  grade 1: 38,0-39,0 Cº; grade 2: >39,0-40,0 Cº; grade 3: >40,0 Cº for ≤ 24 hours; grade 4: >40,0 Cº for > 24 hours

SECONDARY OUTCOMES:
OSDI questionnaire | 4 months after treatment
  Change in severity of dry eye symptoms as assessed with the OSDI questionnaire with a score of 0-100, where 0 is "no symptoms" and 100 is "severe symptoms"
Schirmer's I test | 4 months after treatment
  Change in tear production as evaluated with the Schirmer's I test
Tear osmolarity | 4 months after treatment
  Change in tear osmolarity measured with TearLab(TM)
Ocular SICCA Grading Score | 4 months after treatment
  Change in objective signs of DED as evaluated with the Ocular SICCA Grading Score from 0-12 where 0 is "no staining of the ocular surface" and 12 is "severe staining of the ocular surface"
HLA anti-bodies | 4 months after treatment
  Development of anti-HLA anti-bodies evaluated with Luminex HLA anti-body screening

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Heegaard, MD, DMSc, Study Chair — Department of Ophthalmology, Rigshospitalet-Glostrup, University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No